CLINICAL TRIAL: NCT02083185
Title: A Phase 2, Randomized, Open-label, Parallel Group Study to Evaluate the Safety and Efficacy of the Oral GnRH Antagonist TAK-385, Together With a Leuprorelin Observational Cohort, in Patients With Prostate Cancer
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of TAK-385, Together With a Leuprorelin Observational Cohort, in Participants With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C27002; U1111-1162-5028 (Registry Identifier: WHO); 172837 (Registry Identifier: HC-CTD)
Record Dates: First submitted 2014-03-06; First posted 2014-03-11 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: Drug therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Relugolix 80 mg (Experimental): Relugolix 320 mg (loading dose), tablets, orally, on Day 1 followed by relugolix 80 mg, tablets, orally, once daily for 48 weeks plus an optional 48 week extension at the investigator's discretion.
  Interventions: Drug: Relugolix
- Relugolix 120 mg (Experimental): Relugolix 320 mg (loading dose), tablets, orally, on Day 1 followed by relugolix 120 mg, tablets, orally, once daily for 48 weeks plus an optional 48 week extension at the investigator's discretion.
  Interventions: Drug: Relugolix
- Leuprorelin 22.5 mg (Active Comparator): Leuprorelin 22.5 mg, subcutaneous, injection on Day 1 and every 12 Weeks for up to 4 injections (48 weeks).
  Interventions: Drug: Leuprorelin

INTERVENTIONS:
Drug: Relugolix — Relugolix tablets
  Other Names: TAK-835
  Arms: Relugolix 120 mg; Relugolix 80 mg
Drug: Leuprorelin — Leuprorelin subcutaneous injection
  Arms: Leuprorelin 22.5 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy of TAK 385 for achieving and maintaining testosterone suppression (<50 ng/dL).

DETAILED DESCRIPTION:
The drug being tested in this study is called relugolix (TAK-385). Relugolix is being tested to treat people who have prostate cancer. This study will look at achieving and maintaining testosterone suppression (<50 ng/dL).

The study enrolled 136 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Relugolix 80 mg
* Relugolix 120 mg
* Leuprorelin 22.5 mg

Relugolix was administered starting with a 320 mg (loading dose), followed by relugolix 80 mg or 120 mg tablets, for 48 weeks plus an optional 48-week extension at the investigator's discretion. Patients randomized to leuprorelin were administered 22.5 mg subcutaneously on Day 1 and every 12 weeks for 4 injections.

This multicenter trial was conducted in the United States and Canada. The overall time to participate in this study was 114.4 weeks. Participants made multiple visits to the clinic and at 12 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria

Each participant must meet all of the following inclusion criteria to be enrolled in the study:

1. Male participant 18 years or older.
2. Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma.
3. Candidate for androgen deprivation therapy (ADT) for the management of hormone-sensitive prostate cancer with 1 of the following clinical disease states: 1) advanced localized disease not suitable for primary therapy, 2) evidence of prostate-specific antigen (PSA) biochemical or clinical relapse following primary surgery or radiation therapy of curative intent, or 3) newly diagnosed metastatic disease that is asymptomatic or not threatening to vital organs.
4. Appropriate serum testosterone and serum PSA concentration at screening as specified in the protocol.
5. A body mass index (BMI) ≥ 18.0 at screening and/or baseline.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening and/or baseline.
7. Male participants, even if surgically sterilized, who agree to practice effective barrier contraception or agree to practice true abstinence.
8. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
9. Suitable venous access for the study-required blood sampling, including pharmacokinetic (PK) and pharmacodynamic (PD) Sampling.

Exclusion Criteria

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

1. In participants with advanced, localized M0N1 or M1 disease, the presence of clinically significant symptoms or threat to vital organs requiring immediate gonadotropin-releasing hormone (GnRH) /combined or complete androgen blockade (CAB) therapy, chemotherapy, or radiotherapy.
2. Previously received androgen deprivation therapy (ADT) for more than 8 months total duration (if ADT was received for 8 months or less, then that ADT must have been completed at least 2 years prior to screening).
3. Visceral metastases (liver or lung).
4. Features of the participant's medical condition that may make ADT unnecessary or not indicated.
5. Scheduled for additional surgical or (salvage) radiation therapy within 6 months after baseline evaluations.
6. History of surgical castration.
7. Diagnosis of or treatment for another malignancy within the 2 years before the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
8. Abnormal screening and/or baseline laboratory values as specified in the protocol.
9. History of any significant cardiac condition within 6 months before receiving the first dose of study drug.
10. Electrocardiogram (ECG) abnormalities as specified in the protocol
11. Congenital long QT syndrome.
12. Current use of Class IA (e.g., quinidine, procainamide) or Class III (e.g., amiodarone, sotalol) antiarrhythmic medications.
13. Uncontrolled hypertension despite appropriate medical therapy. Participants may be re-screened after referral and further management of hypertension.
14. Known, previously diagnosed human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life-threatening illness unrelated to prostate cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study. Specific screening for chronic viral illness is at the discretion of the site and/or local institutional review board (IRB).
15. Treatment with any investigational products within 3 months before the first dose of study drug.
16. A primary family member (spouse, parent, child, or sibling of the participant) is involved in the conduct of the study or is a study site employee.
17. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-385, including difficulty swallowing tablets.
18. Use of any medication, or food products listed in the excluded medications and dietary products table within 2 weeks before the first dose of study drug. Participant must have no history of amiodarone use in the 6 months before the first dose of TAK-385.
19. Admission or evidence of alcohol or drug abuse or use of illicit drugs.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 136 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (23):
- United States (19):
  - Birmingham, Alabama
  - San Diego, California
  - Denver, Colorado
  - Daytona Beach, Florida
  - Jeffersonville, Indiana
  - Wichita, Kansas
  - Shreveport, Louisiana
  - Omaha, Nebraska
  - Lawrenceville, New Jersey
  - Garden City, New York
  - Syracuse, New York
  - Cincinnati, Ohio
  - Springfield, Oregon
  - Lancaster, Pennsylvania
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Virginia Beach, Virginia
- Canada (4):
  - Abbotsford, British Columbia
  - Vancouver, British Columbia
  - Montreal, Quebec
  - Québec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in Canada and the United States from 26 March 2014 to 23 February 2017.
Pre-assignment Details: Participants with a diagnosis of prostate cancer were enrolled in 1 of 2 dose levels of TAK-385 (80 or 120 mg) or leuprorelin 22.5 mg.
Groups:
- Relugolix 80 mg: Relugolix 320 mg (loading dose), tablets, orally, on Day 1 followed by relugolix 80 mg, tablets, orally, once daily for 48 weeks plus an optional 48 week extension at the investigator's discretion. Bicalutamide is allowed for firs 4 weeks per investigator's discretion.
- Relugolix 120 mg: Relugolix 320 mg (loading dose), tablets, orally, on Day 1 followed by relugolix 120 mg, tablets, orally, once daily for 48 weeks plus an optional 48 week extension at the investigator's discretion. Bicalutamide is allowed for firs 4 weeks per investigator's discretion.
Period: Overall Study
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Started | 56 | 56 | 24
Safety Population | 56 | 54 | 24
Completed | 36 | 27 | 17
Not Completed | 20 | 29 | 7
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Withdrawal by Subject | 9 | 15 | 1
Not completed — Death | 2 | 2 | 1
Not completed — Reason not Specified | 9 | 6 | 5
Not completed — Study Terminated by Sponsor | 0 | 1 | 0
Not completed — Did not Receive Study Drug | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg | Total
Number analyzed (Participants) | 56 | 54 | 24 | 134
Age, Continuous [Mean (Full Range); unit: years] | 72.3 (9.25) [50 to 91] | 72.1 (8.06) [49 to 87] | 68.3 (6.77) [56 to 82] | 70.9 [49 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 56 | 54 | 24 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 2 | 10
  Not Hispanic or Latino | 51 | 50 | 22 | 123
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 45 | 43 | 24 | 112
  Black or African American | 9 | 10 | 0 | 19
  Asian | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 48 | 23 | 122
  Canada | 5 | 6 | 1 | 12
Height [Mean (Full Range); unit: cm] | 176.92 (8.855) [149.9 to 198.1] | 177.83 (8.459) [157.5 to 198.1] | 177.63 (7.580) [162.6 to 188.0] | 177.46 [149.9 to 198.1]
Weight [Mean (Full Range); unit: kg] | 90.49 (21.632) [56.4 to 193.2] | 92.16 (17.645) [57.3 to 149.5] | 96.10 (17.297) [68.2 to 145.9] | 92.92 [56.4 to 193.2]
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 28.815 (5.9592) [19.51 to 54.66] | 29.077 (4.6509) [18.13 to 39.36] | 30.452 (4.9601) [23.03 to 41.28] | 29.448 [18.13 to 54.66]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Effective Castration Rate Over 24 Weeks
Description: Effective Castration rate is defined as the observed percentage of participants who have testosterone concentrations less than (<) 50 nanogram per deciliter (ng/dL) (1.73 nanomole per liter [nmol/L]) at all scheduled visits beginning after 4 weeks of treatment.
Time Frame: Day 1 of Week 5 to Day 1 of Week 25
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
percentage of participants | 91 [80.4 to 97.0] | 91 [79.7 to 96.9] | 96 [78.9 to 99.9]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Related to Vital Signs
Description: Vital signs included oral temperature, pulse rate, supine systolic and diastolic blood pressure, standing systolic and diastolic blood pressure, and weight. Any TEAEs that were associated with vital signs were reported.
Time Frame: From first dose of study drug to 30 days after last dose of study drug up to 106.7 weeks
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
participants
  Syncope | 3 | 2 | 0
  Hypertension | 1 | 4 | 1
  Hypotension | 1 | 2 | 0
  Arrhythmia | 0 | 1 | 0
  Bradycardia | 2 | 0 | 0
  Tachycardia | 1 | 1 | 1
  Heart rate irregular | 1 | 0 | 0
  Weight increased | 4 | 2 | 0
  Weight decreased | 1 | 0 | 2
  Pyrexia | 3 | 0 | 0

3. Secondary Outcome: Number of Participants With TEAEs Related to Physical Examination
Description: Physical examination consists of examinations of the following body systems: (1) eyes; (2) ears, nose, throat; (3) cardiovascular system; (4) respiratory system; (5) gastrointestinal system; (6) dermatologic system; (7) extremities; (8) musculoskeletal system; (9) nervous system; (10) lymph nodes; and (11) physical examinations other than body systems described in (1) to (10) including slit lamp examination of the anterior eye. Any TEAEs Related to physical examination were reported.
Time Frame: From first dose of study drug to 30 days after last dose of study drug up to 106.7 weeks
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
participants
  Weight increased | 4 | 2 | 0
  Weight decreased | 1 | 0 | 2
  Ophthalmological examination abnormal | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With TEAEs Related to 12-lead Electrocardiogram (ECG) Findings
Description: A single 12-lead ECG was performed. ECGs were read and interpreted locally and reviewed if indicated by the study monitor. ECG abnormalities were reported as AEs.
Time Frame: From first dose of study drug to 30 days after last dose of study drug up to 106.7 weeks
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With TEAES Related to Clinical Laboratory Test Results
Description: Abnormal clinical laboratory values (serum chemistry and hematology) were reported as AEs if they were considered by the investigator to be a clinically significant change from Baseline or led to premature discontinuation of study treatment, dose modification, or other therapeutic intervention.
Time Frame: From first dose of study drug to 30 days after last dose of study drug up to 106.7 weeks
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
participants
  Alanine aminotransferase increased | 7 | 3 | 4
  Aspartate aminotransferase increased | 6 | 1 | 3
  Gamma-glutamyltransferase increased | 3 | 1 | 2
  Blood triglycerides increased | 3 | 0 | 1
  Blood bilirubin increased | 1 | 0 | 0
  Hepatic enzyme increased | 0 | 1 | 0
  Prostatic specific antigen increased | 1 | 1 | 1
  Blood cholesterol increased | 0 | 2 | 0
  Low density lipoprotein increased | 1 | 0 | 0
  Blood glucose increased | 1 | 1 | 0
  Glycosylated haemoglobin increased | 0 | 1 | 0
  Blood creatinine increased | 0 | 1 | 0
  Blood lactate dehydrogenase increased | 2 | 0 | 0
  Blood alkaline phosphatase increased | 1 | 0 | 0
  Blood phosphorus increased | 1 | 0 | 0
  Blood potassium increased | 1 | 0 | 0
  Blood thyroid stimulating hormone increased | 0 | 1 | 0
  Blood testosterone increased | 0 | 0 | 1

6. Secondary Outcome: Number of Participants Reporting One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A SAE is any AE that results in death, is life threatening, requires hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event.
Time Frame: From first dose of study drug to 30 days after last dose of study drug up to 106.7 weeks
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
participants
  Any Adverse Event | 53 | 53 | 23
  SAEs | 10 | 7 | 2

7. Secondary Outcome: Percentage of Participants With Prostate-Specific Antigen (PSA) Response of ≥ 50% and ≥ 90% Reduction at 4 Weeks
Description: PSA Response is defined as a reduction in PSA from Baseline and is reported for 2 categories: ≥ 50% reduction and ≥ 90% reduction.
Time Frame: Week 5, Day 1
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
percentage of participants
  ≥ 50% PSA reduction | 75 | 83 | 17
  ≥ 90% PSA reduction | 13 | 6 | 0

8. Secondary Outcome: Prostate-Specific Antigen Nadir
Description: PSA nadir is the lowest PSA achieved after treatment.
Time Frame: During Weeks 1 to 24
Population: Safety population included all randomized participants who received at least 1 dose of study drug. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per liter (µg/L)
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 54 | 53 | 24
micrograms per liter (µg/L) | 1.8 (7.20) | 5.2 (26.15) | 0.6 (1.03)

9. Secondary Outcome: Serum Prostate-Specific Antigen Concentration at the End of Weeks 12 and 24
Description: Blood was collected and serum concentrations of PSA were obtained using a validated laboratory test at a central laboratory facility.
Time Frame: Day 1 of Weeks 13 and 25
Population: Safety population included all randomized participants who received at least 1 dose of study drug. Here 'n' is the number of participants analyzed at the specific timepoint.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
μg/L
  Week 13, Day 1: number analyzed (Participants) | 53 | 53 | 24
  Week 13, Day 1 | 2.651 (10.0624) | 5.786 (26.4243) | 0.916 (1.4478)
  Week 25, Day 1: number analyzed (Participants) | 50 | 50 | 23
  Week 25, Day 1 | 1.936 (7.5731) | 2.360 (7.3103) | 0.624 (1.0693)

10. Secondary Outcome: Time to Achieve Testosterone Concentrations < 50 ng/dL and < 20 ng/dL
Time Frame: During Weeks 1 to 24
Population: Safety population included all randomized participants who received at least 1 dose of study drug. If a participant has all post first dose testosterone measurements >= 50 ng/dL, the participant's time to castration was censored at the last testosterone measurement that is >= 50 ng/dL.
Measure: Median (Full Range); unit: days
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
days
  Time to Castration (< 50 ng/dL) | 4 [4 to 106] | 4 [4 to 57] | 29 [15 to 57]
  Time to Profound Castration (< 20 ng/dL) | 15 [4 to 141] | 15 [4 to 189] | 29 [15 to 113]

11. Secondary Outcome: TAK-385 Plasma Concentrations
Time Frame: Day 1 of Weeks 1, 2, 3, 5, 9, 13, 17, 25, 37, 49 pre-dose; Day 4 of Week 1 pre-dose; Day 1 of Weeks 5, 13, 2 hrs post-dose
Population: Safety population included all randomized participants who received at least 1 dose of study drug (TAK-835). Here 'n' is the number of participants analyzed at the specific timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Relugolix 80 mg | Relugolix 120 mg
Number analyzed (Participants) | 56 | 54
nanograms per milliliter (ng/mL)
  Week 1, Day 1 pre-dose: number analyzed (Participants) | 51 | 54
  Week 1, Day 1 pre-dose | 0 (0) | 0 (0)
  Week 1, Day 4 pre-dose: number analyzed (Participants) | 51 | 52
  Week 1, Day 4 pre-dose | 9.9 (13.63) | 14.2 (18.52)
  Week 2, Day 1 pre-dose: number analyzed (Participants) | 54 | 53
  Week 2, Day 1 pre-dose | 6.3 (6.32) | 8.7 (10.10)
  Week 3, Day 1 pre-dose: number analyzed (Participants) | 55 | 54
  Week 3, Day 1 pre-dose | 5.4 (3.24) | 10.3 (14.77)
  Week 5, Day 1 pre-dose: number analyzed (Participants) | 52 | 54
  Week 5, Day 1 pre-dose | 5.2 (2.79) | 8.4 (9.85)
  Week 5, Day 1, 2 hours post-dose: number analyzed (Participants) | 51 | 52
  Week 5, Day 1, 2 hours post-dose | 25.3 (21.76) | 45.4 (42.67)
  Week 9, Day 1 pre-dose: number analyzed (Participants) | 50 | 52
  Week 9, Day 1 pre-dose | 4.9 (3.47) | 8.0 (5.82)
  Week 13, Day 1 pre-dose: number analyzed (Participants) | 53 | 53
  Week 13, Day 1 pre-dose | 5.5 (3.39) | 9.0 (7.15)
  Week 13, Day 1, 2 hours post-dose: number analyzed (Participants) | 51 | 50
  Week 13, Day 1, 2 hours post-dose | 24.1 (23.16) | 42.2 (37.04)
  Week 17, Day 1 pre-dose: number analyzed (Participants) | 50 | 52
  Week 17, Day 1 pre-dose | 6.3 (8.12) | 8.9 (6.80)
  Week 25, Day 1 pre-dose: number analyzed (Participants) | 50 | 49
  Week 25, Day 1 pre-dose | 7.3 (11.07) | 11.5 (14.15)
  Week 37, Day 1 pre-dose: number analyzed (Participants) | 44 | 45
  Week 37, Day 1 pre-dose | 6.3 (7.29) | 10.9 (16.94)
  Week 49, Day 1 pre-dose: number analyzed (Participants) | 45 | 39
  Week 49, Day 1 pre-dose | 5.9 (4.98) | 9.4 (8.32)

12. Secondary Outcome: Serum Luteinizing Hormone (LH) Concentrations
Description: Blood was collected and serum concentrations of LH in milli international units per milliliters (mIU/mL) were obtained using a validated laboratory test at a central laboratory facility.
Time Frame: Baseline and Day 4 of Week 1, Day 1 of Weeks 2, 3, 5,13, 25 and 49, End of Treatment (EOT - 106.4 Weeks), Follow-up (110.4 Weeks) and End of Study (114.4 Weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
mIU/mL
  Week 1, Day 4: number analyzed (Participants) | 54 | 52 | 22
  Week 1, Day 4 | 0.665 (0.6982) | 0.595 (0.5467) | 17.551 (13.1433)
  Week 2, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Week 2, Day 1 | 0.548 (0.6683) | 0.638 (1.3988) | 8.279 (5.8986)
  Week 3, Day 1: number analyzed (Participants) | 54 | 53 | 22
  Week 3, Day 1 | 0.341 (0.5851) | 0.388 (0.7887) | 3.171 (2.7636)
  Week 5, Day 1: number analyzed (Participants) | 54 | 53 | 24
  Week 5, Day 1 | 0.424 (1.4941) | 0.203 (0.3580) | 0.508 (0.4327)
  Week 13, Day 1: number analyzed (Participants) | 52 | 51 | 24
  Week 13, Day 1 | 0.229 (0.6003) | 0.183 (0.2542) | 0.277 (0.8253)
  Week 25, Day 1: number analyzed (Participants) | 49 | 49 | 23
  Week 25, Day 1 | 0.195 (0.2524) | 0.175 (0.1365) | 0.134 (0.0992)
  Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 20
  Week 49, Day 1 | 0.341 (0.3948) | 0.288 (0.2479) | 0.138 (0.1677)
  EOT: number analyzed (Participants) | 42 | 45 | 18
  EOT | 3.189 (3.6928) | 2.704 (2.5312) | 0.585 (1.6775)
  Follow-Up: number analyzed (Participants) | 23 | 23 | 15
  Follow-Up | 8.624 (5.3685) | 9.510 (5.2926) | 0.525 (1.0187)
  End of Study: number analyzed (Participants) | 40 | 31 | 16
  End of Study | 7.182 (8.0509) | 9.306 (7.9054) | 1.394 (1.7702)

13. Secondary Outcome: Serum Follicle Stimulating Hormone (FSH) Concentrations
Description: Blood was collected and serum concentrations of FSH were obtained using a validated laboratory test at a central laboratory facility.
Time Frame: Day 1 of Weeks 2, 5, 13, 25, 49, EOT (106.4 Weeks), Follow-up (110.4 Weeks) and End of Study (114.4 Weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
IU/L
  Week 2, Day 1: number analyzed (Participants) | 52 | 52 | 22
  Week 2, Day 1 | 3.112 (3.0612) | 3.183 (2.8956) | 7.650 (5.4542)
  Week 5, Day 1: number analyzed (Participants) | 54 | 52 | 24
  Week 5, Day 1 | 1.248 (2.6737) | 1.035 (1.0479) | 2.946 (1.4428)
  Week 13, Day 1: number analyzed (Participants) | 52 | 50 | 24
  Week 13, Day 1 | 1.137 (2.4242) | 0.908 (0.8104) | 4.625 (2.5594)
  Week 25, Day 1: number analyzed (Participants) | 49 | 48 | 23
  Week 25, Day 1 | 1.090 (0.9932) | 1.344 (0.9675) | 5.043 (2.8221)
  Week 49, Day 1: number analyzed (Participants) | 46 | 42 | 20
  Week 49, Day 1 | 1.802 (1.3956) | 1.938 (1.2169) | 5.145 (2.8201)
  EOT: number analyzed (Participants) | 31 | 22 | 2
  EOT | 5.377 (4.1261) | 5.691 (2.9528) | 5.250 (3.0406)
  Follow-Up: number analyzed (Participants) | 15 | 10 | 1
  Follow-Up | 16.160 (11.0517) | 14.610 (6.1553) | 9.200 (0)
  End of Study: number analyzed (Participants) | 39 | 28 | 14
  End of Study | 11.441 (8.7613) | 15.768 (12.3329) | 5.943 (3.6185)

14. Secondary Outcome: Serum Sex Hormone-binding Globulin (SHBG) Concentrations
Description: Blood was collected and serum concentrations of SHBG were obtained using a validated laboratory test at a central laboratory facility.
Time Frame: Day 1 of Weeks 2, 5, 13, 25, 49, EOT (106.4 Weeks), Follow-up (110.4 Weeks) and End of Study (114.4 Weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
nanomoles per liter (nmol/L)
  Week 2, Day 1: number analyzed (Participants) | 54 | 51 | 24
  Week 2, Day 1 | 50.811 (15.8822) | 48.594 (17.7492) | 39.029 (16.8910)
  Week 5, Day 1: number analyzed (Participants) | 54 | 54 | 22
  Week 5, Day 1 | 49.641 (16.7048) | 49.185 (21.1707) | 43.786 (20.0484)
  Week 13, Day 1: number analyzed (Participants) | 52 | 52 | 24
  Week 13, Day 1 | 49.210 (19.3704) | 50.538 (23.2109) | 41.858 (18.1416)
  Week 25, Day 1: number analyzed (Participants) | 50 | 50 | 23
  Week 25, Day 1 | 47.998 (18.8690) | 50.774 (23.3292) | 40.839 (16.3732)
  Week 49, Day 1: number analyzed (Participants) | 46 | 41 | 21
  Week 49, Day 1 | 50.607 (18.0377) | 54.022 (26.1070) | 38.237 (18.6708)
  EOT: number analyzed (Participants) | 31 | 22 | 1
  EOT | 50.013 (21.5189) | 54.105 (20.8439) | 23.000 (0)
  Follow-Up: number analyzed (Participants) | 15 | 10 | 0
  Follow-Up | 45.433 (14.7416) | 60.250 (28.1206) |
  End of Study: number analyzed (Participants) | 39 | 30 | 14
  End of Study | 51.103 (17.8497) | 51.063 (23.1018) | 39.014 (13.1876)

15. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-P25 Score
Description: EORTC QLQ-PR25 is an EORTC module designed to supplement the QLQ-C30 for any application in prostate cancer consisting of 25 questions distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Questions use are answered using a 4-point scale: 1=Not at all to 4 =Very much. All raw domain scores are linearly transformed to a 0 to 100 scale, with higher scores reflecting either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of activity or functioning (sexual). A positive change from Baseline in activity or functioning scales and negative change from Baseline in symptom scales indicates improvement.
Time Frame: Baseline and Day 1 of Weeks 5,13, 25, 37 and 49, EOT (106.4 Weeks), Follow-up (110.4 Weeks) and End of Study (114.4 Weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
score on a scale
  Sexual Activity: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Sexual Activity: Week 5, Day 1 | -6.0 (29.25) | -14.4 (22.39) | -7.6 (20.25)
  Sexual Activity: Week 13, Day 1: number analyzed (Participants) | 50 | 51 | 24
  Sexual Activity: Week 13, Day 1 | -9.3 (18.49) | -17.3 (27.28) | -11.1 (19.45)
  Sexual Activity: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Sexual Activity: Week 25, Day 1 | -9.4 (25.24) | -19.8 (31.82) | -18.8 (20.90)
  Sexual Activity: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 21
  Sexual Activity: Week 37, Day 1 | -12.0 (27.81) | -14.4 (31.70) | -14.3 (21.27)
  Sexual Activity: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Sexual Activity: Week 49, Day 1 | -13.0 (28.40) | -19.1 (36.24) | -17.5 (31.39)
  Sexual Activity: EOT: number analyzed (Participants) | 35 | 35 | 13
  Sexual Activity: EOT | -15.7 (18.05) | -18.1 (43.79) | -30.8 (27.09)
  Sexual Activity: Follow-up: number analyzed (Participants) | 20 | 29 | 14
  Sexual Activity: Follow-up | -9.2 (18.32) | -24.6 (32.09) | -14.3 (34.50)
  Sexual Activity: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Sexual Activity: End of Study | -7.9 (25.04) | -15.5 (35.89) | -21.9 (24.13)
  Sexual Functioning: Week 5, Day 1: number analyzed (Participants) | 21 | 17 | 12
  Sexual Functioning: Week 5, Day 1 | -9.9 (24.53) | -2.0 (29.25) | -4.2 (14.43)
  Sexual Functioning: Week 13, Day 1: number analyzed (Participants) | 15 | 12 | 10
  Sexual Functioning: Week 13, Day 1 | -8.3 (20.89) | -1.4 (29.27) | 0.8 (27.34)
  Sexual Functioning: Week 25, Day 1: number analyzed (Participants) | 16 | 12 | 7
  Sexual Functioning: Week 25, Day 1 | -4.7 (22.97) | -12.5 (33.80) | -16.7 (23.07)
  Sexual Functioning: Week 37, Day 1: number analyzed (Participants) | 14 | 13 | 8
  Sexual Functioning: Week 37, Day 1 | -10.7 (18.90) | -12.8 (17.55) | -19.8 (17.22)
  Sexual Functioning: Week 49, Day 1: number analyzed (Participants) | 12 | 9 | 7
  Sexual Functioning: Week 49, Day 1 | -16.7 (23.84) | -13.9 (27.95) | 6.0 (23.43)
  Sexual Functioning: EOT: number analyzed (Participants) | 8 | 7 | 2
  Sexual Functioning: EOT | -16.7 (25.97) | -10.7 (6.30) | 37.5 (53.03)
  Sexual Functioning: Follow-up: number analyzed (Participants) | 8 | 4 | 4
  Sexual Functioning: Follow-up | 3.1 (21.33) | -10.4 (18.48) | 2.1 (73.40)
  Sexual Functioning: End of Study: number analyzed (Participants) | 13 | 10 | 3
  Sexual Functioning: End of Study | -11.5 (22.70) | -4.2 (21.96) | -13.9 (12.73)
  Urinary Symptoms: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Urinary Symptoms: Week 5, Day 1 | 2.0 (12.60) | 1.8 (7.84) | 4.2 (7.57)
  Urinary Symptoms: Week 13, Day 1: number analyzed (Participants) | 50 | 51 | 24
  Urinary Symptoms: Week 13, Day 1 | 1.9 (11.64) | 3.8 (7.54) | 6.8 (10.70)
  Urinary Symptoms: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Urinary Symptoms: Week 25, Day 1 | 3.6 (15.46) | 5.1 (12.28) | 7.2 (10.60)
  Urinary Symptoms: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 21
  Urinary Symptoms: Week 37, Day 1 | 3.4 (14.89) | 4.2 (10.24) | 12.9 (14.61)
  Urinary Symptoms: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Urinary Symptoms: Week 49, Day 1 | 4.0 (11.98) | 6.5 (11.18) | 9.9 (11.45)
  Urinary Symptoms: EOT: number analyzed (Participants) | 35 | 35 | 13
  Urinary Symptoms: EOT | 3.3 (14.00) | 7.1 (13.35) | 9.0 (12.83)
  Urinary Symptoms: Follow-up: number analyzed (Participants) | 20 | 19 | 14
  Urinary Symptoms: Follow-up | -1.0 (11.30) | 5.9 (14.52) | 9.8 (7.42)
  Urinary Symptoms: End of study: number analyzed (Participants) | 36 | 29 | 16
  Urinary Symptoms: End of study | 2.2 (10.84) | 4.5 (14.04) | 6.8 (13.08)
  Bowel Symptoms: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Bowel Symptoms: Week 5, Day 1 | 1.9 (7.24) | 1.1 (6.81) | 0.3 (5.75)
  Bowel Symptoms: Week 13, Day 1: number analyzed (Participants) | 50 | 51 | 24
  Bowel Symptoms: Week 13, Day 1 | 1.0 (4.95) | 1.8 (8.55) | 2.4 (7.57)
  Bowel Symptoms: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Bowel Symptoms: Week 25, Day 1 | 3.1 (7.22) | 0.3 (6.87) | 1.1 (4.57)
  Bowel Symptoms: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 21
  Bowel Symptoms: Week 37, Day 1 | 3.8 (7.80) | 1.5 (7.60) | 3.2 (7.21)
  Bowel Symptoms: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Bowel Symptoms: Week 49, Day 1 | 3.0 (6.44) | 0.0 (6.97) | 2.4 (7.04)
  Bowel Symptoms: EOT: number analyzed (Participants) | 35 | 35 | 13
  Bowel Symptoms: EOT | 2.1 (6.18) | 2.4 (7.98) | 2.6 (6.26)
  Bowel Symptoms: Follow-up: number analyzed (Participants) | 20 | 19 | 14
  Bowel Symptoms: Follow-up | 0.0 (4.68) | 2.2 (9.95) | 2.4 (8.91)
  Bowel Symptoms: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Bowel Symptoms: End of Study | 2.1 (5.03) | -0.3 (6.49) | 1.0 (9.56)
  HTRS: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  HTRS: Week 5, Day 1 | 5.6 (8.98) | 5.0 (8.03) | 3.5 (8.94)
  HTRS: Week 13, Day 1: number analyzed (Participants) | 50 | 51 | 24
  HTRS: Week 13, Day 1 | 9.2 (9.95) | 10.8 (10.80) | 7.2 (9.48)
  HTRS: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  HTRS: Week 25, Day 1 | 11.7 (10.07) | 11.3 (11.40) | 10.9 (9.98)
  HTRS: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 21
  HTRS: Week 37, Day 1 | 13.3 (10.51) | 12.2 (13.17) | 13.2 (13.32)
  HTRS: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  HTRS: Week 49, Day 1 | 14.4 (12.39) | 9.6 (11.04) | 15.9 (12.82)
  HTRS: EOT: number analyzed (Participants) | 35 | 35 | 13
  HTRS: EOT | 12.9 (12.33) | 14.0 (16.13) | 17.9 (12.25)
  HTRS: Follow-up: number analyzed (Participants) | 20 | 19 | 14
  HTRS: Follow-up | 7.5 (8.51) | 6.1 (9.05) | 15.9 (15.69)
  HTRS: End of Study: number analyzed (Participants) | 36 | 29 | 16
  HTRS: End of Study | 10.8 (11.03) | 9.8 (11.27) | 12.5 (12.75)
  Incontinence Aid: Week 5, Day 1: number analyzed (Participants) | 20 | 18 | 4
  Incontinence Aid: Week 5, Day 1 | 0.0 (21.63) | -1.9 (17.98) | -16.7 (19.25)
  Incontinence Aid: Week 13, Day 1: number analyzed (Participants) | 19 | 19 | 4
  Incontinence Aid: Week 13, Day 1 | 0.0 (22.22) | -1.8 (13.49) | -16.7 (19.25)
  Incontinence Aid: Week 25, Day 1: number analyzed (Participants) | 19 | 19 | 2
  Incontinence Aid: Week 25, Day 1 | 3.5 (21.93) | 0.0 (15.71) | -16.7 (23.57)
  Incontinence Aid: Week 37, Day 1: number analyzed (Participants) | 16 | 19 | 2
  Incontinence Aid: Week 37, Day 1 | 8.3 (25.82) | -1.8 (13.49) | -16.7 (23.57)
  Incontinence Aid: Week 49, Day 1: number analyzed (Participants) | 19 | 15 | 3
  Incontinence Aid: Week 49, Day 1 | 7.0 (23.78) | -2.2 (15.26) | -22.2 (19.25)
  Incontinence Aid: EOT: number analyzed (Participants) | 11 | 11 | 2
  Incontinence Aid: EOT | 6.1 (20.10) | 6.1 (20.10) | -16.7 (23.57)
  Incontinence Aid: Follow-up: number analyzed (Participants) | 6 | 8 | 1
  Incontinence Aid: Follow-up | 0.0 (21.08) | -8.3 (15.43) | -33.3 (0)
  Incontinence Aid: End of Study: number analyzed (Participants) | 12 | 14 | 1
  Incontinence Aid: End of Study | 0.0 (20.10) | -4.8 (22.10) | -33.3 (0)

16. Secondary Outcome: Percent Change From Baseline of Aging Male Survey (AMS) Total Score
Description: AMS scale is a self-administered questionnaire used to: 1) assess symptoms of aging (independent from those that are disease related) between groups of males under different conditions; 2) evaluate the severity of symptoms over time; and 3) measure changes before and after androgen therapy. Each question was answered between 1=none to 5=extremely severe for 17 items from psychological (5 items), somatic (7 items), and sexual (5 items) categories. Total score is sum of all the item scores and range from 17 (minimum) to 85 (maximum), where high score indicated high level of symptoms.
Time Frame: as for outcome 15
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
percent change
  Week 5, Day 1: number analyzed (Participants) | 54 | 52 | 24
  Week 5, Day 1 | 3.914 (24.4749) | 10.872 (29.6532) | 10.083 (27.1933)
  Week 13, Day 1: number analyzed (Participants) | 52 | 51 | 24
  Week 13, Day 1 | 14.781 (24.0185) | 17.259 (33.9921) | 21.887 (36.5551)
  Week 25, Day 1: number analyzed (Participants) | 49 | 48 | 23
  Week 25, Day 1 | 20.272 (35.2952) | 20.353 (34.2105) | 46.995 (55.3558)
  Week 37, Day 1: number analyzed (Participants) | 47 | 46 | 22
  Week 37, Day 1 | 24.136 (33.8595) | 24.466 (35.6742) | 49.422 (61.1264)
  Week 49, Day 1: number analyzed (Participants) | 46 | 41 | 21
  Week 49, Day 1 | 30.122 (38.1093) | 24.377 (33.6078) | 59.971 (60.3579)
  EOT: number analyzed (Participants) | 36 | 35 | 13
  EOT | 18.857 (37.9260) | 28.644 (35.6470) | 60.952 (63.3615)
  Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Follow-Up | 15.754 (21.8158) | 13.031 (33.7754) | 53.834 (61.6683)
  End of Study: number analyzed (Participants) | 37 | 29 | 16
  End of Study | 16.270 (24.2582) | 21.304 (46.0184) | 49.879 (54.1540)

17. Secondary Outcome: Change From Baseline in EORTC QLQ-C30
Description: The EORTC QLQ-C30 included 30 questions comprising 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, nausea/vomiting), single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties) and a global health and QOL scale. Most questions used a 4-point scale (1=Not at all to 4=Very much); 2 questions used a 7-point scale (1= Very poor to 7=Excellent). All domain scores were calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem. A positive change from Baseline in quality og life or functioning scales and negative change from Baseline in symptom or difficulties scales indicates improvement.
Time Frame: Day 1 of Weeks 5, 13, 25, 37, 49, 73, 97, EOT (106.4 Weeks), Follow-up (110.4 Weeks) and End of Study (114.4 Weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Number analyzed (Participants) | 56 | 54 | 24
score on a scale
  Quality of Life: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Quality of Life: Week 5, Day 1 | -2.7 (14.51) | -4.0 (17.50) | -5.2 (13.64)
  Quality of Life: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Quality of Life: Week 13, Day 1 | -2.3 (15.37) | -2.0 (14.87) | -7.3 (15.21)
  Quality of Life: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Quality of Life: Week 25, Day 1 | -6.4 (20.21) | -2.3 (15.45) | -6.9 (16.98)
  Quality of Life: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Quality of Life: Week 37, Day 1 | -6.0 (20.69) | -7.4 (20.58) | -11.7 (18.84)
  Quality of Life: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Quality of Life: Week 49, Day 1 | -7.2 (19.18) | -7.3 (18.18) | -8.3 (17.87)
  Quality of Life: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Quality of Life: Week 73, Day 1 | -3.4 (17.18) | -12.0 (13.19) |
  Quality of Life: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Quality of Life: Week 97, Day 1 | -6.6 (20.71) | -2.2 (18.18) |
  Quality of Life: EOT: number analyzed (Participants) | 35 | 35 | 13
  Quality of Life: EOT | -4.8 (16.82) | -7.1 (15.80) | -13.5 (24.19)
  Quality of Life: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Quality of Life: Follow-Up | -5.4 (12.17) | -8.8 (22.13) | -13.7 (19.50)
  Quality of Life: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Quality of Life: End of Study | -7.9 (18.14) | -10.1 (15.49) | -10.9 (13.85)
  Physical Functioning: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Physical Functioning: Week 5, Day 1 | 0.9 (9.87) | -0.9 (7.70) | -0.8 (8.41)
  Physical Functioning: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Physical Functioning: Week 13, Day 1 | 0.3 (9.23) | -4.4 (8.50) | -0.3 (14.77)
  Physical Functioning: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Physical Functioning: Week 25, Day 1 | -2.8 (15.24) | -5.3 (10.20) | -2.0 (14.42)
  Physical Functioning: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Physical Functioning: Week 37, Day 1 | -4.8 (13.60) | -6.2 (12.26) | -4.2 (16.78)
  Physical Functioning: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Physical Functioning: Week 49, Day 1 | -4.3 (13.79) | -5.2 (9.95) | -7.0 (17.32)
  Physical Functioning: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Physical Functioning: Week 73, Day 1 | -5.1 (9.20) | -8.5 (8.72) |
  Physical Functioning: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Physical Functioning: Week 97, Day 1 | -8.1 (9.58) | -6.0 (8.86) |
  Physical Functioning: EOT: number analyzed (Participants) | 35 | 35 | 13
  Physical Functioning: EOT | -3.4 (15.37) | -9.3 (14.66) | -2.6 (22.20)
  Physical Functioning: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Physical Functioning: Follow-Up | -4.0 (9.02) | -6.3 (19.18) | -3.8 (21.52)
  Physical Functioning: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Physical Functioning: End of Study | -8.9 (13.52) | -9.0 (13.48) | -2.9 (20.22)
  Role Functioning: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Role Functioning: Week 5, Day 1 | 0.3 (14.43) | -0.3 (15.30) | 2.8 (8.03)
  Role Functioning: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Role Functioning: Week 13, Day 1 | -1.0 (17.13) | -3.6 (16.09) | 1.4 (21.93)
  Role Functioning: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Role Functioning: Week 25, Day 1 | -4.9 (21.18) | -6.3 (19.03) | -2.2 (23.19)
  Role Functioning: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Role Functioning: Week 37, Day 1 | -10.9 (23.10) | -10.0 (16.82) | -4.5 (24.22)
  Role Functioning: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Role Functioning: Week 49, Day 1 | -8.1 (23.20) | -8.9 (22.70) | -7.1 (19.42)
  Role Functioning: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Role Functioning: Week 73, Day 1 | -8.0 (13.08) | -6.7 (14.43) |
  Role Functioning: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Role Functioning: Week 97, Day 1 | -8.8 (15.08) | -4.4 (12.22) |
  Role Functioning: EOT: number analyzed (Participants) | 35 | 35 | 13
  Role Functioning: EOT | -9.5 (21.88) | -8.6 (20.76) | -5.1 (29.17)
  Role Functioning: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Role Functioning: Follow-Up | -10.0 (16.58) | -10.5 (31.04) | -7.1 (29.75)
  Role Functioning: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Role Functioning: End of Study | -10.6 (12.69) | -13.2 (21.99) | -1.0 (26.15)
  Emotional Functioning: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Emotional Functioning: Week 5, Day 1 | 1.9 (8.59) | 0.3 (12.45) | 1.7 (10.98)
  Emotional Functioning: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Emotional Functioning: Week 13, Day 1 | -0.7 (11.53) | -1.1 (12.70) | -1.4 (12.69)
  Emotional Functioning: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Emotional Functioning: Week 37, Day 1 | -4.3 (12.26) | -1.7 (11.73) | -9.8 (20.35)
  Emotional Functioning: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Emotional Functioning: Week 49, Day 1 | -3.0 (14.01) | -1.4 (12.06) | -4.4 (18.56)
  Emotional Functioning: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Emotional Functioning: Week 73, Day 1 | -2.0 (9.36) | -2.3 (16.578) |
  Emotional Functioning: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Emotional Functioning: Week 97, Day 1 | -2.6 (12.44) | 2.6 (7.88) |
  Emotional Functioning: EOT: number analyzed (Participants) | 35 | 35 | 13
  Emotional Functioning: EOT | -3.6 (11.30) | -7.4 (17.12) | -14.1 (24.15)
  Emotional Functioning: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Emotional Functioning: Follow-Up | -3.3 (8.72) | -1.3 (19.50) | -8.9 (23.22)
  Emotional Functioning: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Emotional Functioning: End of Study | -5.3 (12.62) | -0.6 (14.42) | -8.3 (17.74)
  Cognitive Functioning: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Cognitive Functioning: Week 5, Day 1 | -0.9 (11.97) | -4.2 (14.71) | -2.8 (10.62)
  Cognitive Functioning: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Cognitive Functioning: Week 13, Day 1 | -1.0 (13.50) | -7.5 (16.44) | -5.6 (16.05)
  Cognitive Functioning: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Cognitive Functioning: Week 25, Day 1 | -0.7 (14.16) | -3.8 (15.08) | -2.9 (11.95)
  Cognitive Functioning: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Cognitive Functioning: Week 37, Day 1 | -5.8 (12.28) | -5.6 (16.67) | -9.8 (15.99)
  Cognitive Functioning: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Cognitive Functioning: Week 49, Day 1 | -2.6 (12.29) | -6.1 (13.82) | -11.9 (16.79)
  Cognitive Functioning: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Cognitive Functioning: Week 73, Day 1 | -5.7 (15.61) | -7.3 (13.68) |
  Cognitive Functioning: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Cognitive Functioning: Week 97, Day 1 | -6.1 (8.26) | -7.0 (13.96) |
  Cognitive Functioning: EOT: number analyzed (Participants) | 20 | 29 | 14
  Cognitive Functioning: EOT | -2.9 (14.84) | -10.0 (23.64) | -12.8 (21.68)
  Cognitive Functioning: Follow-Up: number analyzed (Participants) | 20 | 29 | 14
  Cognitive Functioning: Follow-Up | -0.8 (14.78) | -7.0 (21.74) | -10.7 (15.48)
  Cognitive Functioning: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Cognitive Functioning: End of Study | -2.3 (16.01) | -7.5 (18.14) | -3.1 (16.35)
  Social Functioning: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Social Functioning: Week 5, Day 1 | 0.3 (16.50) | -1.3 (14.33) | 4.2 (16.48)
  Social Functioning: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Social Functioning: Week 13, Day 1 | 1.6 (13.85) | -3.3 (12.48) | -0.7 (18.04)
  Social Functioning: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Social Functioning: Week 25, Day 1 | -1.0 (16.98) | -6.3 (20.23) | -202 (22.08)
  Social Functioning: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Social Functioning: Week 37, Day 1 | -2.5 (18.58) | -5.9 (16.34) | -7.6 (20.40)
  Social Functioning: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Social Functioning: Week 49, Day 1 | -3.7 (15.85) | -9.8 (20.74) | -8.7 (26.15)
  Social Functioning: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Social Functioning: Week 73, Day 1 | -2.9 (11.84) | -6.0 (15.12) |
  Social Functioning: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Social Functioning: Week 97, Day 1 | -5.3 (15.77) | -4.4 (14.53) |
  Social Functioning: EOT: number analyzed (Participants) | 35 | 35 | 13
  Social Functioning: EOT | -5.2 (16.55) | -10.0 (21.08) | -6.4 (30.84)
  Social Functioning: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Social Functioning: Follow-Up | -3.3 (10.26) | -8.8 (25.07) | -4.8 (22.10)
  Social Functioning: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Social Functioning: End of Study | -3.7 (16.48) | -9.2 (19.20) | 0.0 (14.91)
  Fatigue: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Fatigue: Week 5, Day 1 | 1.9 (13.74) | 4.3 (14.95) | 3.2 (15.19)
  Fatigue: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Fatigue: Week 13, Day 1 | 6.1 (17.40) | 8.9 (15.72) | 8.3 (11.47)
  Fatigue: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Fatigue: Week 25, Day 1 | 6.3 (21.12) | 13.2 (15.66) | 13.5 (18.94)
  Fatigue: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Fatigue: Week 37, Day 1 | 9.7 (21.55) | 14.1 (19.30) | 16.7 (21.89)
  Fatigue: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Fatigue: Week 49, Day 1 | 10.9 (24.33) | 11.1 (16.67) | 20.1 (23.47)
  Fatigue: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Fatigue: Week 73, Day 1 | 10.0 (24.19) | 14.7 (13.88) |
  Fatigue: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Fatigue: Week 97, Day 1 | 5.8 (22.94) | 9.9 (18.48) |
  Fatigue: EOT: number analyzed (Participants) | 35 | 35 | 13
  Fatigue: EOT | 12.1 (27.53) | 15.9 (20.22) | 20.5 (18.62)
  Fatigue: Follow-up: number analyzed (Participants) | 20 | 19 | 14
  Fatigue: Follow-up | 7.2 (15.41) | 6.4 (19.71) | 13.5 (21.87)
  Fatigue: End of study: number analyzed (Participants) | 36 | 29 | 16
  Fatigue: End of study | 11.4 (17.72) | 12.3 (22.88) | 8.3 (19.25)
  Nausea and Vomiting: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Nausea and Vomiting: Week 5, Day 1 | -1.3 (6.41) | 0.6 (9.88) | 3.5 (6.91)
  Nausea and Vomiting: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Nausea and Vomiting: Week 13, Day 1 | 0.7 (7.42) | 0.7 (7.42) | 1.4 (4.71)
  Nausea and Vomiting: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Nausea and Vomiting: Week 25, Day 1 | 0.0 (9.10) | 0.0 (3.44) | 2.9 (6.46)
  Nausea and Vomiting: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Nausea and Vomiting: Week 37, Day 1 | 0.4 (8.95) | 1.1 (7.45) | 4.5 (9.17)
  Nausea and Vomiting: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Nausea and Vomiting: Week 49, Day 1 | -1.9 (7.30) | 0.8 (6.40) | 4.8 (11.95)
  Nausea and Vomiting: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Nausea and Vomiting: Week 73, Day 1 | 0.0 (4.45) | 0.7 (3.33) |
  Nausea and Vomiting: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Nausea and Vomiting: Week 97, Day 1 | 5.3 (14.75) | 1.8 (9.45) |
  Nausea and Vomiting: Week EOT: number analyzed (Participants) | 35 | 35 | 13
  Nausea and Vomiting: Week EOT | -0.5 (8.56) | 1.9 (8.83) | 7.7 (14.62)
  Nausea and Vomiting: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Nausea and Vomiting: Follow-Up | 3.3 (16.75) | 0.9 (3.82) | 0.0 (6.54)
  Nausea and Vomiting: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Nausea and Vomiting: End of Study | 1.4 (9.24) | -1.1 (4.30) | 0.0 (6.09)
  Pain: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Pain: Week 5, Day 1 | -1.6 (16.75) | 0.6 (16.82) | 3.5 (18.38)
  Pain: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Pain: Week 13, Day 1 | -1.0 (17.77) | 3.3 (18.86) | 4.2 (26.12)
  Pain: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Pain: Week 25, Day 1 | 0.3 (22.67) | 2.8 (16.61) | 2.9 (22.84)
  Pain: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Pain: Week 37, Day 1 | 2.9 (23.65) | 5.9 (21.37) | 11.4 (34.27)
  Pain: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Pain: Week 49, Day 1 | 3.3 (23.19) | 6.5 (18.59) | 7.9 (31.46)
  Pain: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Pain: Week 73, Day 1 | 6.9 (18.64) | 7.3 (14.50) |
  Pain: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Pain: Week 97, Day 1 | 5.3 (19.29) | 0.0 (14.70) |
  Pain: EOT: number analyzed (Participants) | 35 | 35 | 13
  Pain: EOT | -0.5 (25.08) | 6.7 (24.32) | 6.4 (35.05)
  Pain: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Pain: Follow-Up | 9.2 (21.95) | 10.5 (23.05) | 1.2 (28.84)
  Pain: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Pain: End of Study | 6.5 (17.03) | 6.9 (19.17) | -2.1 (30.96)
  Dyspnea: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Dyspnea: Week 5, Day 1 | -0.6 (21.17) | 2.6 (17.27) | 5.6 (18.82)
  Dyspnea: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Dyspnea: Week 13, Day 1 | 5.9 (22.81) | 6.5 (21.10) | 8.3 (20.26)
  Dyspnea: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Dyspnea: Week 25, Day 1 | 4.2 (26.30) | 8.3 (22.28) | 8.7 (22.96)
  Dyspnea: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Dyspnea: Week 37, Day 1 | 6.5 (21.80) | 11.1 (22.47) | 22.7 (26.00)
  Dyspnea: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Dyspnea: Week 49, Day 1 | 6.7 (22.02) | 9.8 (20.06) | 17.5 (30.95)
  Dyspnea: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Dyspnea: Week 73, Day 1 | 8.0 (19.22) | 9.3 (18.05) |
  Dyspnea: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Dyspnea: Week 97, Day 1 | 10.5 (19.41) | 8.8 (18.73) |
  Dyspnea: EOT: number analyzed (Participants) | 35 | 35 | 13
  Dyspnea: EOT | 7.6 (24.37) | 14.3 (20.27) | 20.5 (32.03)
  Dyspnea: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Dyspnea: Follow-Up | 11.7 (22.36) | 8.8 (26.86) | 14.3 (25.20)
  Dyspnea: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Dyspnea: End of Study | 11.1 (19.52) | 14.9 (26.10) | 8.3 (31.03)
  Insomnia: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Insomnia: Week 5, Day 1 | -1.3 (24.43) | 3.2 (17.79) | 1.4 (18.33)
  Insomnia: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Insomnia: Week 13, Day 1 | 2.6 (20.92) | 9.8 (21.39) | 6.9 (19.61)
  Insomnia: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Insomnia: Week 25, Day 1 | 6.3 (30.49) | 12.5 (24.43) | 8.7 (22.96)
  Insomnia: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Insomnia: Week 37, Day 1 | 2.2 (24.75) | 8.1 (22.65) | 18.2 (32.08)
  Insomnia: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Insomnia: Week 49, Day 1 | 6.7 (29.81) | 7.3 (22.99) | 6.3 (32.69)
  Insomnia: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Insomnia: Week 73, Day 1 | 2.3 (33.25) | 10.7 (23.01) |
  Insomnia: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Insomnia: Week 97, Day 1 | 10.5 (27.34) | 10.5 (19.41) |
  Insomnia: EOT: number analyzed (Participants) | 35 | 35 | 13
  Insomnia: EOT | 6.7 (35.97) | 7.6 (26.92) | 7.7 (24.17)
  Insomnia: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Insomnia: Follow-Up | 5.0 (19.57) | 0.0 (27.22) | 4.8 (25.68)
  Insomnia: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Insomnia: End of Study | 1.9 (28.67) | 5.7 (21.95) | 10.4 (29.11)
  Appetite Loss: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Appetite Loss: Week 5, Day 1 | -3.8 (14.11) | 0.6 (21.38) | 2.8 (13.61)
  Appetite Loss: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Appetite Loss: Week 13, Day 1 | -0.7 (18.25) | -0.7 (20.54) | 0.0 (13.90)
  Appetite Loss: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Appetite Loss: Week 25, Day 1 | -3.5 (19.74) | 0.0 (19.45) | 2.9 (17.15)
  Appetite Loss: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Appetite Loss: Week 37, Day 1 | -0.7 (17.90) | 2.2 (16.51) | 0.0 (14.55)
  Appetite Loss: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Appetite Loss: Week 49, Day 1 | -0.7 (16.65) | 0.8 (15.79) | 4.8 (15.94)
  Appetite Loss: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Appetite Loss: Week 73, Day 1 | -2.3 (12.38) | 5.3 (18.46) |
  Appetite Loss: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Appetite Loss: Week 97, Day 1 | 0.0 (15.71) | 3.5 (15.29) |
  Appetite Loss: EOT: number analyzed (Participants) | 35 | 35 | 13
  Appetite Loss: EOT | -3.8 (15.70) | 8.6 (16.85) | 2.6 (16.45)
  Appetite Loss: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Appetite Loss: Follow-Up | 0.0 (15.29) | 3.5 (18.90) | -2.4 (15.82)
  Appetite Loss: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Appetite Loss: End of Study | -1.9 (13.67) | 3.4 (13.64) | 0.0 (24.34)
  Constipation: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Constipation: Week 5, Day 1 | 0.6 (20.14) | 1.9 (17.97) | 1.4 (6.80)
  Constipation: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Constipation: Week 13, Day 1 | 3.9 (21.75) | 5.2 (19.29) | 5.6 (12.69)
  Constipation: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Constipation: Week 25, Day 1 | 2.8 (19.25) | 6.3 (25.41) | 1.4 (15.82)
  Constipation: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Constipation: Week 37, Day 1 | 5.8 (20.25) | 8.1 (26.74) | 1.5 (12.50)
  Constipation: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Constipation: Week 49, Day 1 | 2.2 (19.33) | 7.3 (20.43) | 1.6 (7.27)
  Constipation: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Constipation: Week 73, Day 1 | 1.1 (18.86) | 1.3 (17.95) |
  Constipation: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Constipation: Week 97, Day 1 | 1.8 (26.00) | 3.5 (21.93) |
  Constipation: EOT: number analyzed (Participants) | 35 | 35 | 13
  Constipation: EOT | 3.8 (22.54) | 1.9 (17.97) | 0.0 (13.61)
  Constipation: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Constipation: Follow-Up | 5.0 (24.84) | 10.5 (24.98) | 0.0 (13.07)
  Constipation: End Of Study: number analyzed (Participants) | 36 | 29 | 16
  Constipation: End Of Study | 3.7 (19.15) | 5.7 (17.97) | 0.0 (17.21)
  Diarrhea: Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Diarrhea: Week 5, Day 1 | -1.9 (12.08) | 1.9 (13.87) | 1.4 (11.95)
  Diarrhea: Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Diarrhea: Week 13, Day 1 | 3.9 (18.44) | 2.0 (23.49) | 0.0 (9.83)
  Diarrhea: Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Diarrhea: Week 25, Day 1 | 2.8 (17.97) | 5.6 (19.85) | 2.9 (13.90)
  Diarrhea: Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Diarrhea: Week 37, Day 1 | 3.6 (17.54) | 0.7 (15.06) | 6.1 (13.16)
  Diarrhea: Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Diarrhea: Week 49, Day 1 | 3.0 (17.15) | -1.6 (16.59) | 1.6 (16.59)
  Diarrhea: Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Diarrhea: Week 73, Day 1 | 4.6 (17.19) | 1.3 (15.15) |
  Diarrhea: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Diarrhea: Week 97, Day 1 | 7.0 (17.84) | 0.0 (15.71) |
  Diarrhea: EOT: number analyzed (Participants) | 35 | 35 | 13
  Diarrhea: EOT | 4.8 (14.33) | 2.9 (16.90) | 5.1 (18.49)
  Diarrhea: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Diarrhea: Follow-Up | 3.3 (10.26) | 0.0 (19.25) | 4.8 (12.10)
  Diarrhea: End Of Study: number analyzed (Participants) | 36 | 29 | 16
  Diarrhea: End Of Study | 1.9 (17.72) | -1.1 (18.86) | 2.1 (19.12)
  Financial Difficulties:Week 5, Day 1: number analyzed (Participants) | 53 | 52 | 24
  Financial Difficulties:Week 5, Day 1 | -1.3 (9.16) | 2.6 (21.74) | -1.4 (18.33)
  Financial Difficulties:Week 13, Day 1: number analyzed (Participants) | 51 | 51 | 24
  Financial Difficulties:Week 13, Day 1 | -2.0 (16.88) | -0.7 (20.54) | 2.8 (23.91)
  Financial Difficulties:Week 25, Day 1: number analyzed (Participants) | 48 | 48 | 23
  Financial Difficulties:Week 25, Day 1 | -3.5 (12.38) | 0.7 (20.03) | 4.3 (23.15)
  Financial Difficulties:Week 37, Day 1: number analyzed (Participants) | 46 | 45 | 22
  Financial Difficulties:Week 37, Day 1 | -2.9 (19.66) | 1.5 (18.74) | 7.6 (20.40)
  Financial Difficulties:Week 49, Day 1: number analyzed (Participants) | 45 | 41 | 21
  Financial Difficulties:Week 49, Day 1 | -5.2 (20.04) | 0.8 (18.99) | 3.2 (17.97)
  Financial Difficulties:Week 73, Day 1: number analyzed (Participants) | 29 | 25 | 0
  Financial Difficulties:Week 73, Day 1 | 0.0 (8.91) | 2.7 (16.44) |
  Financial Difficulties: Week 97, Day 1: number analyzed (Participants) | 19 | 19 | 0
  Financial Difficulties: Week 97, Day 1 | 5.3 (20.07) | 1.8 (20.71) |
  Financial Difficulties: EOT: number analyzed (Participants) | 35 | 35 | 13
  Financial Difficulties: EOT | -3.8 (19.42) | 5.7 (20.59) | 2.6 (16.45)
  Financial Difficulties: Follow-Up: number analyzed (Participants) | 20 | 19 | 14
  Financial Difficulties: Follow-Up | 5.0 (12.21) | 1.8 (20.71) | 11.9 (33.61)
  Financial Difficulties: End of Study: number analyzed (Participants) | 36 | 29 | 16
  Financial Difficulties: End of Study | -2.8 (18.47) | 3.4 (22.44) | 0.0 (21.08)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after last dose of study drug up to 106.7 weeks
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Relugolix 80 mg | Relugolix 120 mg | Leuprorelin 22.5 mg
Serious Adverse Events (participants affected / at risk) | 10/56 | 7/54 | 2/24
Other Adverse Events (participants affected / at risk) | 53/56 | 50/54 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix 80 mg (N=56) | Relugolix 120 mg (N=54) | Leuprorelin 22.5 mg (N=24)
Bradycardia (Cardiac disorders) | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with leuprorelin 22.5 mg and is not related.
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with relugolix 80 mg and is not related.
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with relugolix 80 mg is not related.
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with relugolix 120 mg and is not related.
Sudden death (General disorders) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with relugolix 120 mg and is not related.
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix 80 mg (N=56) | Relugolix 120 mg (N=54) | Leuprorelin 22.5 mg (N=24)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 3
Hot flush (Vascular disorders) | 32 | 35 | 15
Hypertension (Vascular disorders) | 1 | 4 | 1
Fatigue (General disorders) | 11 | 19 | 7
Pyrexia (General disorders) | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 4 | 5 | 1
Urinary tract infection (Infections and infestations) | 5 | 2 | 1
Sinusitis (Infections and infestations) | 3 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 3 | 0
Cataract (Eye disorders) | 7 | 13 | 0
Visual acuity reduced (Eye disorders) | 2 | 4 | 0
Dry eye (Eye disorders) | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 7 | 3 | 4
Aspartate aminotransferase increased (Investigations) | 6 | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 1 | 2
Weight increased (Investigations) | 4 | 2 | 0
Blood triglycerides increased (Investigations) | 3 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 0
Insomnia (Psychiatric disorders) | 1 | 5 | 2
Libido decreased (Psychiatric disorders) | 1 | 3 | 1
Depression (Psychiatric disorders) | 1 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Dizziness (Nervous system disorders) | 2 | 4 | 0
Headache (Nervous system disorders) | 2 | 3 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0
Gynaecomastia (Reproductive system and breast disorders) | 3 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 3
Corneal dystrophy (Congenital, familial and genetic disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.